CLINICAL TRIAL: NCT05908552
Title: A Novel Non-Opioid Topical Therapy for Chronic Musculoskeletal Pain
Brief Title: Topical Cannabis for Chronic Musculoskeletal Pain
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 22-1289; 25B2360 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2023-01-17; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Chronic Pain; Musculoskeletal Pain; Joint Pain
Keywords: topical; cannabis
MeSH Terms: conditions — Chronic Pain; Musculoskeletal Pain; Arthralgia; Marijuana Abuse

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Our proposal objective is to evaluate if state-regulated topical CBD-based products relieve chronic musculoskeletal pain and/or absorb into the bloodstream.

DETAILED DESCRIPTION:
The goal of this study is to learn more about the analgesic efficacy of state-regulated topical cannabinoid products (creams, lotions, salves, etc) and to determine if these topical products are absorbed systemically and can be detected in blood samples. Given that state-regulated dispensary products cannot be brought onto the university campus, this observational study design utilizes a Mobile Pharmacology Laboratory that will go to study participants' homes. Blood samples and other assessments will taken in the mobile lab prior to use of a topical cannabinoid product and at several time points afterwards (4 hours, 24 hours, and 2 weeks). Participants will also collect microsamples of blood using a small device at home at three time points during the first 2-72 hours after application of the product.

ELIGIBILITY:
Some inclusion/exclusion criteria are purposely omitted at this time to preserve scientific integrity. They will be included after the trial is complete.

Inclusion Criteria:

* Chronic peripheral joint pain
* Desire and intent to use a topical cannabinoid product containing cannabidiol (CBD) or a combination of CBD and tetrahydrocannabinol (THC) to alleviate this pain

Exclusion Criteria:

* Current or prior use of topical cannabis
* Unwilling or unable to discontinue other (non-topical) cannabis use for four weeks prior to and during study participation through week two
* Intent to use a THC-predominant topical product (ratio greater than 1:1 of THC to CBD)
* Current or history of substance use disorder
* History or diagnosis of schizophrenia, bipolar or a psychotic disorder
* Surgery on the affected musculoskeletal location within the 3 months prior to enrollment
* Planned surgery or procedure on the affected musculoskeletal location during participation in the study
* Allergy or prior severe adverse reaction to cannabis (cardiovascular event, psychosis, etc)
* Current or prior cannabis abuse/dependence
* Cognitive disability that interferes with ability to provide consent or understand study procedures
* History of seizure disorder
* Pending legal action or workers compensation
* Pregnant females or females intending to become pregnant during the study period
* Lactating females
* Chronic/severe medical illness (renal disease, liver disease, cancer, significant cardiovascular disease, or history of myocardial infarction)
* Active component military

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with chronic pain of the peripheral joints (such as knee, ankle, and shoulder) who are interested in initiating use of a topical cannabinoid will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in in PROMIS Pain Interference Score from Baseline to 2 months | Assessed at baseline, 4 hours, 24 hours, 2 weeks and 2 months
  The PROMIS Pain Interference (Short Form 6a) includes 6 items that assess the self-reported consequences of pain on various aspects of life including social, cognitive, emotional, physical and recreational activities. Participants rate these consequences on a Likert Scale that ranges from 1 (Not at all) to 5 (Very much). The scores are then converted to T-scores, with higher values indicating greater pain interference.
Levels of plasma cannabinoid and cannabinoid metabolites | Baseline to 2 weeks
  Four venous blood samples will be obtained at baseline, 4 hours, 24 hours, and 2 weeks after first use of the selected topical cannabinoid.

SECONDARY OUTCOMES:
Opioid and non-opioid pain medications use | Daily through 2 weeks
  Participant self-report of opioid and non-opioid analgesic use
Reported drug effects | Baseline, 4 hours, 24 hours, 2 weeks, 2 months
  Subjective ratings of psychoactive effects ("high,'' ''impaired,'' ''stoned,'' ''like the drug effect,'' ''sedated,'' ''confused,'' ''nauseated,'' ''desire more of the drug,'' ''anxious,'' ''down,'' ''hungry,'') measured on a 100-mm VAS
Change in in PROMIS Pain Intensity Score from Baseline to 2 months | Assessed at baseline, 4 hours, 24 hours, 2 weeks and 2 months
  The PROMIS Pain Intensity (Short Form 3a) includes 3 items that assess how much a person hurts. The first two items assess pain intensity using a 7-day recall period (items include the phrase "the past 7 days") while the last item asks patients to rate their pain intensity "right now." Participants rate their pain on a Likert Scale that ranges from: 1 (Had no pain) to 5 (Very severe).
Change in Patient-Reported Outcomes Measurement Information System (PROMIS)-29 Profile from Baseline to 2 months | Assessed at baseline, 4 hours, 24 hours, 2 weeks and 2 months
  The PROMIS-29 Profile assesses physiological, social, and psychological outcomes using a comprehensive set of biopsychosocial domains. These domains include physical function, anxiety, depression, fatigue, sleep, ability to participate in social roles and/or activities, pain interference, and pain intensity. The questionnaire responses are ranked on a 5-point Likert Scale, and pain intensity is rated on an 11-point scale. Higher scores reflect a greater presence of the measured domain. For symptom-oriented domains (anxiety, depression, fatigue, pain interference, and sleep disturbance), higher scores indicate more severe symptomatology, while for function-oriented domains (physical functioning and social role), higher scores indicate better functioning. For instance, a high sleep disturbance score indicates significant levels of sleep disruption, whereas a high physical functioning score indicates better physical capabilities.
Change in Patients' Global Impression of Change (PGIC) from Baseline to 2 Months | Assessed at baseline, 4 hours, 24 hours, 2 weeks and 2 months
  The Patient Global Impression of Change (PGIC) is a self-report measure used in chronic pain clinical trials to assess a patient's perception of treatment efficacy. The PGIC uses a 7-point scale where patients rate their overall improvement, ranging from "very much improved" to "very much worse."
Change Patient Specific Functional Scale from Baseline to 2 Months | Assessed at baseline, 4 hours, 24 hours, 2 weeks and 2 months
  The Patient Specific Functional Scale is an 11-point scale where "0" represents "unable to perform activity" and "10" represents "Able to perform activity at the same level as before injury or problem". Participants rate their ability to perform up to five important activities that they find difficult due to their musculoskeletal pain.
Change in NIH Toolbox® List Sorting Working Memory Test from Baseline to 2 Weeks | Assessed at baseline, 4 hours, 24 hours, 2 weeks
  Test of working memory - the capacity of an individual to hold information in a short-term buffer and manipulate the information. All cognitive data will be represented by raw scores and T scores. We will assess changes over time in patients comparing their 4 hour, 24 hour, 2 week time-points to baseline.
Change in NIH Toolbox® Oral Symbol Digit Test from Baseline to 2 Weeks | Assessed at baseline, 4 hours, 24 hours, 2 weeks
  Test of processing speed - the amount of time it takes to mentally process a set amount of information, or the amount of information that can be processed within a certain unit of time. It is a measure that reflects mental efficiency. All cognitive data will be represented by raw scores and T scores. We will assess changes over time in patients comparing their 4 hour, 24 hour, 2 week time-points to baseline.
Change in NIH Toolbox® Flanker Inhibitory Control and Attention Test from Baseline to 2 Weeks | Assessed at baseline, 4 hours, 24 hours, 2 weeks
  Test of executive function - the capacity to plan, organize and monitor the execution of behaviors that are strategically directed in a goal-oriented manner) and attention (allocation of one's limited capacities to deal with an abundance of environmental stimulation) test. All cognitive data will be represented by raw scores and T scores. We will assess changes over time in patients comparing their 4 hour, 24 hour, 2 week time-points to baseline.
Change in NIH Toolbox® Pattern Comparison Processing Speed Test from Baseline to 2 Weeks | Assessed at baseline, 4 hours, 24 hours, 2 weeks
  Test of processing speed - the amount of time it takes to mentally process a set amount of information, or the amount of information that can be processed within a certain unit of time. It is a measure that reflects mental efficiency. All cognitive data will be represented by raw scores and T scores. We will assess changes over time in patients comparing their 4 hour, 24 hour, 2 week time-points to baseline.
Change in NIH Toolbox® Picture Vocabulary Test from Baseline to 2 Weeks | Assessed at baseline, 4 hours, 24 hours, 2 weeks
  Test of vocabulary knowledge. All cognitive data will be represented by raw scores and T scores. We will assess changes over time in patients comparing their 4 hour, 24 hour, 2 week time-points to baseline.
Change in Fine Motor Function from Baseline to 2 Weeks | Assessed at baseline, 4 hours, 24 hours, 2 weeks
  The Grooved Pegboard Test will be used to test fine motor function. The manipulative dexterity test described in the protocol consists of a board with twenty-five holes containing randomly positioned slots and pegs. The pegs have a key along one side and must be rotated to match the corresponding hole before insertion. This test evaluates the speed of performance in a fine motor task and assesses both sides of the body.
Change in Gross Motor Function from Baseline to 2 Weeks | Assessed at baseline, 4 hours, 24 hours, 2 weeks
  Change in Gross Motor Function will be assessed by the DRiving Under the Influence of Drugs (DRUID)® tests and Components of the Field Sobriety Tests, including One-Leg Stand, Walk-and-Turn, Modified Romberg Balance. The DRUID® tests measure impairment based on performance of various tasks. Scores range from 0-100, where lower scores indicate better performance. ≥13-point change (from baseline) on DRUID global impairment score = "impaired"; <13-point change (from baseline) = "not impaired". Two or more clues noted during the field sobriety tests indicate impairment.
Abuse liability | Assessed at baseline, 4 hours, 24 hours, 2 weeks and 2 months
  Craving visual analog scale (VAS): Assesses craving for topical cannabinoid on a 100mm visual scale. Drug Effects Questionnaire (DEQ): Assesses the strength of the topical cannabinoid effect
Participant Treatment Expectations and Impressions | Assessed at baseline, 4 hours, 24 hours, 2 weeks and 2 months
  Questionnaires will be conducted to assess participants' treatment expectations and impressions.
Participant Perceived Efficacy | Assessed at baseline, 4 hours, 24 hours, 2 weeks and 2 months
  Questionnaires will be conducted to assess participants' impressions of perceived efficacy of the chosen topical cannabinoid.
Participant Preference vs Other Analgesics | Assessed at baseline, 4 hours, 24 hours, 2 weeks and 2 months
  Questionnaires will be conducted to assess participants' preference for the chosen topical cannabinoid vs other analgesics.
Participant Reported Adverse Effects | Assessed at baseline, 4 hours, 24 hours, 2 weeks and 2 months
  Questionnaires will be conducted to assess participants' reported Adverse Effects
Half life analysis of cannabinoid and cannabinoid metabolites | baseline through 2 weeks
  A total of six blood samples will be obtained and analyzed using population pharmacokinetic modeling with sparse sampling with cannabinoids and their kinetically distinct metabolites.
Clearance analysis of cannabinoid and cannabinoid metabolites | baseline through 2 weeks
  A total of six blood samples will be obtained and analyzed using population pharmacokinetic modeling with sparse sampling with cannabinoids and their kinetically distinct metabolites.
Volume of distribution analysis of cannabinoid and cannabinoid metabolites | baseline through 2 weeks
  A total of six blood samples will be obtained and analyzed using population pharmacokinetic modeling with sparse sampling with cannabinoids and their kinetically distinct metabolites.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Lindley, PhD, Principal Investigator — University of Colorado, Denver; Rachael Rzasa Lynn, MD, Principal Investigator — University of Colorado, Denver

IPD SHARING:
Plan to Share IPD: No